CLINICAL TRIAL: NCT01617681
Title: A 6 Week, Randomized, Multicenter, Double-blind, Double-dummy Study to Evaluate the Dose Response of Valsartan on Blood Pressure Reduction in Children 1-5 Years Old With Hypertension, With or Without Chronic Kidney Disease, Followed by a 20 Week Open-label Titration Phase
Brief Title: Efficacy, Safety and Tolerability of Multiple Doses of Valsartan in Children With Hypertension With or Without CKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAL489K2306; 2011-005991-40 (EudraCT Number)
Record Dates: First submitted 2012-06-06; First posted 2012-06-12 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-08

CONDITIONS: Pediatric Hypertension With or Without CKD
Keywords: Hypertension; CKD; Pediatric
MeSH Terms: conditions — Hypertension | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Valsartan 0.25 mg/kg (Experimental): Valsartan oral solution 0.25mg/kg once daily + matching placebo of valsartan oral solution 4 mg/kg once daily for 6 weeks (period 1)
  Interventions: Drug: VAL489; Drug: VAL489 matching placebo
- Valsartan 4 mg/kg (Experimental): Valsartan oral solution 4 mg/kg once daily + matching placebo of valsartan oral solution 0.25 mg/kg once daily for 6 weeks (period 1)
  Interventions: Drug: VAL489; Drug: VAL489 matching placebo
- Valsartan 1 mg/kg (Experimental): Open-label (Period 2) valsartan will be optionally titrated from 1 mg/kg to 2 mg/kg. Valsartan will continue to be optionally up titrated in 1 mg/kg increments every 4 weeks until maximum dose of 4 mg/kg is achieved. Duration 20 weeks.
  Interventions: Drug: VAL489

INTERVENTIONS:
Drug: VAL489 — Valsartan 3mg/kg oral solution
  Other Names: Diovan
Drug: VAL489 matching placebo — Valsartan 3 mg/kg oral solution
  Other Names: Diovan
  Arms: Valsartan 0.25 mg/kg; Valsartan 4 mg/kg

SUMMARY:
To assess efficacy, safety and tolerability of valsartan when comparing two doses of valsartan in reducing and controlling blood pressure in children with hypertension with or without CKD.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to fulfill all of the following criteria:

Have the ability to provide written informed consent; Have at baseline , a documented diagnosis of hypertension (as defined in the National High Blood Pressure Education Program 2004); MSBP (mean of 3 measurements) must be ≥95th percentile, and ≤25% above the 95th percentile, for age, gender and height, at baseline; CKD patients must be defined as any of the following criteria: Kidney damage for ≥3 months, as defined by structural or functional abnormalities of the kidney, with or without decreased GFR, manifested by one or more of the following features: Abnormalities in the composition of urine, Abnormalities in imaging tests, Abnormalities on kidney biopsy, Estimated eGFR <60 mL/min/1.73m2 for ≥3 months, with or without the other signs of kidney damage described above; Able to swallow the valsartan solution; Body weight must be ≥8 kg and ≤40 kg at baseline; Must be able to safely washout from other antihypertensive therapy (if applicable) Exclusion criteria AST/SGOT or ALT/SGPT >3 times the upper limit of the reference range; Estimated Glomerular Filtration Rate [eGFR] <30 mL/min/1.73m² (calculated using Modified Schwartz Formula); Serum potassium >5.3 mmol/L; Uncontrolled diabetes mellitus, as defined by the investigator; Unilateral, bilateral and graft renal artery stenosis; Current diagnosis of heart failure (NYHA Class II-IV); Patients taking any of the following concomitant medications following screening: RAAS blockers other than study drug, Lithium, Potassium-sparing diuretics, potassium supplements, salt substitutes containing potassium and other substances that may increase potassium levels; Non-steroidal anti-inflammatory drugs (NSAIDS), including selective COX-2 inhibitors, acetylsalicylic acid >3g/day, and non-selective NSAIDs (paracetamol/acetaminophen is permitted); Antidepressant drugs in the class of MAO inhibitors (e.g. phenelzine); Chronic use of stimulant therapy for ADD/ADHD; patients who have coarctation of the aorta with a gradient of ≥30 mmHg; Previous solid organ transplantation except renal transplantation. Renal transplant must have occurred at least 1 year prior to enrollment; Patient must be on stable doses of immunosuppressive therapy and deemed clinically stable by the investigator; Patients known to be positive for the human immunodeficiency virus (HIV) Other protocol defined inclusion/exclusion criteria may apply.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2012-11-08 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2017-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- Belgium (2):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Liège
- Brazil (4):
  - Novartis Investigative Site, Curitibia, Paraná
  - Novartis Investigative Site, Campinas
  - Novartis Investigative Site, Caxias do Sul
  - Novartis Investigative Site, Porto Alegre
- Novartis Investigative Site, Montpellier, France
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Marburg
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Italy (3):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, San Donato Milanese, MI
  - Novartis Investigative Site, Palermo
- Novartis Investigative Site, Vinius, Lithuania
- Poland (8):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Warsaw

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Jankauskiene A, Drozdz D, Wasilewska A, de Paula-Bernardes R, Glazer R, Valentin M, Tan M, Chiang Y, Bapatla K. Efficacy and safety of valsartan in children aged 1-5 years with hypertension, with or without chronic kidney disease: a randomized, double-blind study followed by open-label phase. Curr Med Res Opin. 2021 Dec;37(12):2113-2122. doi: 10.1080/03007995.2021.1982681. Epub 2021 Oct 9. PMID 34543161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 156 patients were screened, of which 127 patients were enrolled in the double blind period 1 of the study. A total of 120 patients (94.5%) completed Period 1 and entered Open Label Period 2.
Pre-assignment Details: Parallel= Period 1 (Double Blind phase) Single= Period 2 (Open Label phase)
Groups:
- CKD Patients Valsartan 0.25 mg/kg: CKD patients: Valsartan oral solution 0.25mg/kg once daily + matching placebo of valsartan oral solution 4 mg/kg once daily for 6 weeks (period 1)
- CKD Patients Valsartan 4 mg/kg: CKD patients: Valsartan oral solution 4 mg/kg once daily + matching placebo of valsartan oral solution 0.25 mg/kg once daily for 6 weeks (period 1)
- Non-CKD Patients Valsartan 0.25 mg/kg: Non-CKD patients: Valsartan oral solution 0.25mg/kg once daily + matching placebo of valsartan oral solution 4 mg/kg once daily for 6 weeks (period 1)
- Non-CKD Patients Valsartan 4 mg/kg: Non-CKD patients: Valsartan oral solution 4 mg/kg once daily + matching placebo of valsartan oral solution 0.25 mg/kg once daily for 6 weeks (period 1)
- Valsartan 1 mg/kg (Period 2): Open-label (Period 2) valsartan will be optionally titrated from 1 mg/kg to 2 mg/kg. Valsartan will continue to be optionally up titrated in 1 mg/kg increments every 4 weeks until maximum dose of 4 mg/kg is achieved. Duration 20 weeks.
Period: Period 1 Double Blind
Arm/Group | CKD Patients Valsartan 0.25 mg/kg | CKD Patients Valsartan 4 mg/kg | Non-CKD Patients Valsartan 0.25 mg/kg | Non-CKD Patients Valsartan 4 mg/kg | Valsartan 1 mg/kg (Period 2)
Started | 32 | 31 | 33 | 31 | 0
Full Analysis Set (FAS) | 31 | 31 | 33 | 31 | 0
Completed | 29 | 30 | 32 | 29 | 0
Not Completed | 3 | 1 | 1 | 2 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0
Period: Period 2 Open Label
Arm/Group | CKD Patients Valsartan 0.25 mg/kg | CKD Patients Valsartan 4 mg/kg | Non-CKD Patients Valsartan 0.25 mg/kg | Non-CKD Patients Valsartan 4 mg/kg | Valsartan 1 mg/kg (Period 2)
Started | 0 | 0 | 0 | 0 | 120
Completed | 0 | 0 | 0 | 0 | 114
Not Completed | 0 | 0 | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CKD Patients Valsartan 0.25 mg/kg | CKD Patients Valsartan 4 mg/kg | Non-CKD Patients Valsartan 0.25 mg/kg | Non-CKD Patients Valsartan 4 mg/kg | Total
Number analyzed (Participants) | 32 | 31 | 33 | 31 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.99 (1.47) | 2.72 (1.33) | 3.7 (1.51) | 3.62 (1.36) | 3.26 (1.466)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 14 | 13 | 47
  Male | 20 | 23 | 19 | 18 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 16 | 14 | 15 | 57
  Not Hispanic or Latino | 20 | 15 | 19 | 16 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Systolic Blood Pressure (MSBP) at Week 6 Endpoint
Description: Patient's blood pressure will be measured in the same position at every visit Systolic and diastolic blood pressures will be measured three times at 2-3 minute intervals. The arithmetic mean of these three blood pressure measurements will be used as the mean office blood pressure (MSBP and MDBP) at Baseline and Week 6 endpoint in Period 1 Double Blind Phase
Time Frame: Baseline, week 6
Population: Full analysis set (FAS) included all randomized patient except for 1 patient that guardian did not sign informed consent
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | CKD Patients Valsartan 0.25 mg/kg | CKD Patients Valsartan 4 mg/kg | Non-CKD Patients Valsartan 0.25 mg/kg | Non-CKD Patients Valsartan 4 mg/kg
Number analyzed (Participants) | 31 | 31 | 33 | 31
mmHg | -1.2 (2.05) | -9.2 (2.05) | -6.9 (1.44) | -7.8 (1.48)
Statistical Analysis 1: Comparison: CKD Patients Valsartan 0.25 mg/kg vs CKD Patients Valsartan 4 mg/kg; Test type: Other; p = 0.0096, ANCOVA; Mean Difference (Net) = -7.9, 95% CI 2-sided [-13.86 to -2.01], Standard Error of Mean 2.96
Statistical Analysis 2: Comparison: Non-CKD Patients Valsartan 0.25 mg/kg vs Non-CKD Patients Valsartan 4 mg/kg; Test type: Other; p = 0.6531, ANCOVA; Mean Difference (Net) = -0.9, 95% CI 2-sided [-5.07 to 3.20], Standard Error of Mean 2.07

2. Secondary Outcome: Change From Baseline in Mean Diastolic Blood Pressure (MDBP) at Week 6
Description: Patient's blood pressure will be measured in the same position at every visit Systolic and diastolic blood pressures will be measured three times at 2-3 minute intervals. The arithmetic mean of these three blood pressure measurements will be used as the mean office blood pressure (MSBP and MDBP) Baseline and Week 6 endpoint in Period 1 Double Blind Phase
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | CKD Patients Valsartan 0.25 mg/kg | CKD Patients Valsartan 4 mg/kg | Non-CKD Patients Valsartan 0.25 mg/kg | Non-CKD Patients Valsartan 4 mg/kg
Number analyzed (Participants) | 31 | 31 | 33 | 31
mmHg | 1.3 (1.79) | -6.5 (1.79) | -1.9 (1.26) | -7.2 (1.30)
Statistical Analysis 1: Comparison: CKD Patients Valsartan 0.25 mg/kg vs CKD Patients Valsartan 4 mg/kg; Test type: Other; p = 0.0030, ANCOVA; Mean Difference (Net) = -7.9, 95% CI 2-sided [-12.94 to -2.78], Standard Error of Mean 2.54
Statistical Analysis 2: Comparison: Non-CKD Patients Valsartan 0.25 mg/kg vs Non-CKD Patients Valsartan 4 mg/kg; Test type: Other; p = 0.0042, ANCOVA; Mean Difference (Net) = -5.4, 95% CI 2-sided [-8.98 to -1.77], Standard Error of Mean 1.80

3. Secondary Outcome: Patients Achieving <90th Percentile for Age, Gender and Height at Week 6 Endpoint in Both MSBP and MDBP
Description: Patient's blood pressure will be measured in the same position at every visit Systolic and diastolic blood pressures will be measured three times at 2-3 minute intervals. The arithmetic mean of these three blood pressure measurements will be used as the mean office blood pressure (MSBP and MDBP) Week 6
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CKD Patients Valsartan 0.25 mg/kg | CKD Patients Valsartan 4 mg/kg | Non-CKD Patients Valsartan 0.25 mg/kg | Non-CKD Patients Valsartan 4 mg/kg
Number analyzed (Participants) | 31 | 31 | 33 | 31
participants | 6 | 9 | 7 | 8
Statistical Analysis 1: Comparison: CKD Patients Valsartan 0.25 mg/kg vs CKD Patients Valsartan 4 mg/kg; Test type: Other; p = 0.411, ANCOVA; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.49 to 5.8]
Statistical Analysis 2: Comparison: Non-CKD Patients Valsartan 0.25 mg/kg vs Non-CKD Patients Valsartan 4 mg/kg; Test type: Other; p = 0.5443, ANCOVA; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.44 to 4.79]

4. Secondary Outcome: CKD Patients Achieving Urine Albumin Creatinine Ratio Percentage Reduction (UACR) >=25% at Week 6
Description: UACR response is defined as percentage change from baseline in UACR≤ 25%. UACR [mg/mmol] = urine albumin [mg/L] / urine creatinine [mmol/L] UACR was collected for CKD patients only. The UACR value at a given visit for a patient was to be derived by the median of the three lab values collected for that visit Week 6.
Time Frame: Week 6 weeks
Population: Full analysis set (FAS) included all randomized patient except for 1 patient that guardian did not sign informed consent - CKD patients only The number of patients with an UACR at baseline and week 6 endpoint (included in the analysis).
Measure: Number; unit: participants
Arm/Group | CKD Patients Valsartan 0.25 mg/kg | CKD Patients Valsartan 4 mg/kg
Number analyzed (Participants) | 27 | 27
participants | 12 | 9
Statistical Analysis 1: Comparison: CKD Patients Valsartan 0.25 mg/kg vs CKD Patients Valsartan 4 mg/kg; Test type: Other; p = 0.2624, ANCOVA; Odds Ratio (OR) = 0.517, 95% CI 2-sided [0.16 to 1.64]

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Groups:
- Valsartan 0.25 mg/kg: All Patients CKD & Non-CKD: Valsartan oral solution 0.25mg/kg once daily + matching placebo of valsartan oral solution 4 mg/kg once daily for 6 weeks (period 1)
- Valsartan 4.0 mg/kg: All Patients CKD & Non-CKD patients: Valsartan oral solution 4 mg/kg once daily + matching placebo of valsartan oral solution 0.25 mg/kg once daily for 6 weeks (period 1)
- All Open Label Patients: Open-label (Period 2) valsartan will be optionally titrated from 1 mg/kg to 2 mg/kg. Valsartan will continue to be optionally up titrated in 1 mg/kg increments every 4 weeks until maximum dose of 4 mg/kg is achieved. Duration 20 weeks.
Arm/Group | Valsartan 0.25 mg/kg | Valsartan 4.0 mg/kg | All Open Label Patients
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/62 | 0/120
Serious Adverse Events (participants affected / at risk) | 2/64 | 2/62 | 6/120
Other Adverse Events (participants affected / at risk) | 19/64 | 13/62 | 62/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan 0.25 mg/kg (N=64) | Valsartan 4.0 mg/kg (N=62) | All Open Label Patients (N=120)
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Mastoiditis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan 0.25 mg/kg (N=64) | Valsartan 4.0 mg/kg (N=62) | All Open Label Patients (N=120)
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 10
Vomiting (Gastrointestinal disorders) | 3 | 1 | 9
Pyrexia (General disorders) | 2 | 3 | 20
Bronchitis (Infections and infestations) | 3 | 0 | 7
Ear infection (Infections and infestations) | 0 | 0 | 7
Nasopharyngitis (Infections and infestations) | 3 | 2 | 9
Respiratory tract infection (Infections and infestations) | 4 | 3 | 6
Tonsillitis (Infections and infestations) | 0 | 2 | 8
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single- site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2012-05-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT01617681/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT01617681/SAP_001.pdf